CLINICAL TRIAL: NCT05261880
Title: Comparison of the Effects of Scaphoid and Hamate Mobilization and Neural Mobilization on Patients With Carpal Tunnel Syndrome: a Randomized Controlled Trial
Brief Title: Comparative Effect of Scaphoid, Hamate Mobilization and Neural Mobilization in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00248
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be single blinded as assessors of the study would be kept blind of the treatment group to which patient will allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization (Experimental): Neural mobilization will be given for 15 minutes with 3 repetitions. After mobilization, Kinesio taping will be applied and it will bandage till the next session.
  Interventions: Other: Neural mobilization
- Scaphoid, hamate mobilization (Experimental): Scaphoid and hamate mobilization for 20 minutes, at the end of session kinesio taping will bandage till the next session.
  Interventions: Other: Scaphoid , hamate mobilization

INTERVENTIONS:
Other: Neural mobilization — Neural mobilization and bone are two common physical therapy interventions used for Carpal Tunnel Syndrome. Neural mobilization reinstates the plasticity of the nervous system and restoring the capacity of stretching.
  Arms: Neural mobilization
Other: Scaphoid , hamate mobilization — Bone mobilization in Carpal Tunnel Syndrome involves gliding at scaphoid and hamate.
  Arms: Scaphoid, hamate mobilization

SUMMARY:
To rule out the effects bone mobilization and neural mobilization in Carpal Tunnel Syndrome.

DETAILED DESCRIPTION:
A Randomized control study of 3 month period will be conducted at Riphah International University Faisalabad. Patients will be enrolled by purposive sampling based on pre-defined inclusion and exclusion criteria. Patients were randomly allocated into groups. The Patients of group A will receive scaphoid, hamate mobilization with kinesio taping and group B will receive neural mobilization with kinesiotaping. Group A will receive neural mobilization and Group B will receive scaphoid and hamate moilization. The Patient's outcome will be distinguished by Visual Analogue scale and the data of the patients will be noted pre-treatment and post-treatment. Informed consent will be taken from each patient. Data entry and analysis will prepare through Statistical Package of Social Sciences Version 20.

ELIGIBILITY:
Inclusion Criteria:

* At median nerve distribution, felt pain and parasthesia Phalen sign positive Tinel sign positive Increase symptoms throughout the night Symptoms that continue for at least 3 weeks

Exclusion Criteria:

* Pregnancy Diabetes Thyroid disease Rheumatoid arthritis Thenar muscle atrophy Weakness of thenar muscle Hand surgery/ bone fracture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 12th Week
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Dynamometer | 12th Week
  It is a small device that the examiner holds against the patient's limb as the patient exerts a maximal force. The examiner counters the force "make test", or tries to break the contraction "break test".
Boston questionnaire | 12th Week
  The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No